CLINICAL TRIAL: NCT00125957
Title: The Effects of Wellbutrin (Bupropion) on Residual and Cognitive Symptoms in SSRI-treated Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Association for Research on Schizophrenia and Affective Disorders. (Unknown)
Responsible Party: Principal Investigator, Beth L. Murphy MD, PhD, Principal Investigator, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005P-000502
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Depression; Major Depressive Disorder; Unipolar Depression
Keywords: depression; serotonin; norepinephrine; SSRI; Wellbutrin; bupropion; executive function; residual symptoms
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depressive Disorder | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wellbutrin first, then Placebo (Experimental): Subjects randomly assigned to the Wellbutrin then Placebo group will receive 100mg BID of Wellbutrin at the first visit following intake (Week 0).Subjects will be increased to 150mg Wellbutrin BID at Week 1 unless moderate/severe side effects are reported. If subject and rater classify 1+ symptom as severe or 2+ symptoms as moderate, subject will continue on 100mg of bupropion qAM. If subject and rater classify 1+ symptom as moderate or 2+ mild as moderate, subject will continue on Wellbutrin 100mg BID. At Week 4, subjects will cross-over to placebo and will continue to take placebo until Week 8.
  Interventions: Drug: Wellbutrin; Drug: Placebo
- Placebo first, then Wellbutrin (Experimental): Subjects randomly assigned to the Placebo then Wellbutrin group will receive placebo until Week 4 when they will cross-over to active drug. At Week 4, subjects will be assigned 100mg Wellbutrin BID. At Week 5, Subjects will be increased to 150mg Wellbutrin BID unless moderate/severe side effects are reported. If subject and rater classify 1+ symptom as severe or 2+ symptoms as moderate, subject will continue on 100mg of Wellbutrin qAM. If subject and rater classify 1+ symptom as moderate or 2+ mild as moderate, subject will continue on bupropion 100mg BID. Subject will continue on the assigned dosage until Week 8 of study.
  Interventions: Drug: Wellbutrin; Drug: Placebo

INTERVENTIONS:
Drug: Wellbutrin
  Other Names: bupropion
Drug: Placebo

SUMMARY:
Many people with depression are treated with a serotonin-specific reuptake inhibitor anti-depressant (SSRI) and feel 'better'. Although many people feel 'better', they do not feel completely 'well'. Often, individuals continue to complain of cognitive problems such as lack of attention, diminished motivation, and impaired problem-solving. This study looks at whether residual and cognitive symptoms of depression in individuals are affected by the addition of Wellbutrin (bupropion).

DETAILED DESCRIPTION:
As many as 65-75% of treated patients continue to experience residual symptoms of depression. Cognitive impairments feature frontal cognitive dysfunction. Many experts believe that executive functions are better predictors of functional level than psychiatric diagnoses.

Frontal cognitive impairment and changes in neuroimaging are seen in individuals depleted of tryptophan, a serotonin precursor. These cognitive changes do not improve following serotonin-specific reuptake inhibitor treatment and at least one study has found that executive dysfunction predicts non-response to fluoxetine. In many patients, remission of mood symptoms in depression requires medications to target non-serotonergic neurotransmitter systems. Brain areas mediating executive functions receive rich noradrenergic inputs, and norepinephrine is known to be intimately involved in many of the executive functions.

A better understanding of serotonergic and catecholaminergic interactions would enable evidence-based treatment of depression which maximizes executive cognitive functions. This study examines the hypothesis that individuals treated with Wellbutrin will have higher scores on tests of executive functions and lower scores on depression indices.

ELIGIBILITY:
Inclusion Criteria:

* Depression
* SSRI-treated

Exclusion Criteria:

* Bipolar disorder
* Serotonin-norepinephrine reuptake inhibitor (SNRI) or bupropion treatment
* Treatment-resistant depression
* Seizure disorder
* Bulimia or anorexia nervosa
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-08; Primary Completion 2010-01 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth L Murphy, MD, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Wellbutrin First, Then Placebo: Subjects randomly assigned to the Wellbutrin first, then Placebo group will receive 100mg BID of Wellbutrin at the first visit following intake (Week 0).Subjects will be increased to 150mg Wellbutrin BID at Week 1 unless moderate/severe side effects are reported. If subject and rater classify 1+ symptom as severe or 2+ symptoms as moderate, subject will continue on 100mg of bupropion qAM. If subject and rater classify 1+ symptom as moderate or 2+ mild as moderate, subject will continue on Wellbutrin 100mg BID. At Week 4, subjects will cross-over to placebo and will continue to take placebo until Week 8.
- Placebo First, Then Wellbutrin: Subjects randomly assigned to the Placebo first, then Wellbutrin group will receive placebo until Week 4 when they will cross-over to active drug. At Week 4, subjects will be assigned 100mg Wellbutrin BID. At Week 5, Subjects will be increased to 150mg Wellbutrin BID unless moderate/severe side effects are reported. If subject and rater classify 1+ symptom as severe or 2+ symptoms as moderate, subject will continue on 100mg of Wellbutrin qAM. If subject and rater classify 1+ symptom as moderate or 2+ mild as moderate, subject will continue on bupropion 100mg BID. Subject will continue on the assigned dosage until Week 8 of study.
Period: First Intervention (3 Weeks)
Arm/Group | Wellbutrin First, Then Placebo | Placebo First, Then Wellbutrin
Started | 15 | 17
Completed | 15 | 17
Not Completed | 0 | 0
Period: Second Intervention (3 Weeks)
Arm/Group | Wellbutrin First, Then Placebo | Placebo First, Then Wellbutrin
Started | 15 | 17
Completed | 15 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Wellbutrin-Placebo: Study subjects randomly assigned to this arm of the study will begin on active drug (100 mg twice daily (BID) of Wellbutrin) at week 1. At week 2, active drug is increased to 150mg BID unless subject reports one or more symptoms that are classified as moderate-severe. At week 4, subjects cross over to placebo for remainder of study. Subjects continue on placebo until end of study at week 8.
- Placebo-Wellbutrin: Subjects randomly assigned to this arm are given placebo at week 1. They will continue on placebo until week 4, at which time they will cross-over to Wellbutrin 100 mg twice daily (BID). At week 5, active drug is increased to 150mg BID unless subject reports one or more symptoms that are classified as moderate-severe. Subjects continue on active drug until end of study at week 8.
- Total: Total of all reporting groups
Arm/Group | Wellbutrin-Placebo | Placebo-Wellbutrin | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Mean (Full Range); unit: years] | 49 [18 to 65] | 47 [22 to 63] | 48 [18 to 65]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 17 | 31
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 6 | 9 | 15
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Median total depression symptoms rating at baseline and follow-up visits. The MADRS consists o 10 questions assessing depression symptoms. All questions are scored on a 0-6 severity scale, with 0 being absent and 4 being most severe. Total scores can range from 0-60.
Time Frame: Baseline and follow-up
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Wellbutrin First, Then Placebo: Subjects randomly assigned to Treatment A will receive Wellbutrin or placebo at Week 1 and will cross over to Wellbutrin or placebo at week 4.
- Placebo First, Then Wellbutrin: Subjects randomly assigned to Treatment B will receive Wellbutrin or placebo at Week 1 and will cross over to Wellbutrin or placebo at week 4.
Arm/Group | Wellbutrin First, Then Placebo | Placebo First, Then Wellbutrin
Number analyzed (Participants) | 15 | 17
units on a scale
  Baseline | 22.0 [19.0 to 24.0] | 18.0 [9.0 to 21.0]
  Follow-up at week 4 | 12.0 [8.0 to 21.0] | 14.0 [5.0 to 19.0]
Statistical Analysis 1: Comparison: Wellbutrin First, Then Placebo vs Placebo First, Then Wellbutrin; Null Hypothesis: There is no difference in the mean change MADRS score between Wellbutrin-Placebo and Placebo-Wellbutrin treatment groups; Test type: Superiority or Other; p = .04, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Hamilton Depression Rating Scale (HAM-D)
Description: Median total depression ratings at baseline and follow-up using the HAM-D. The scale consists of 21 questions that assess depression symptoms. Questions 1-3, 7-11, 15, and 19 are rated on a scale of 0-4, with 0 being not present to and 4 being severe. Questions 4, 5, 12 - 14, 16-18 and 21 are rated from 0-2 with a score of 0 signifying the symptom is absent and a score of 2 as most severe. Item 20 is score on a scale of 0-3 with the same pattern of severity as all other questions. The total score for the HAM-D ranges from 0-63.
Time Frame: Baseline and follow-up
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Wellbutrin First, Then Placebo | Placebo First, Then Wellbutrin
Number analyzed (Participants) | 15 | 17
units on a scale
  Baseline | 21.5 [16 to 29] | 14 [9 to 18]
  Follow-up at week 4 | 13.5 [8 to 17] | 14 [8 to 18]
Statistical Analysis 1: Comparison: Wellbutrin First, Then Placebo vs Placebo First, Then Wellbutrin; Null Hypothesis: There is no difference in the median HAM-D score between Wellbutrin-Placebo and Placebo-Wellbutrin treatment groups; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Groups:
- Bupropion-Placebo: Study subjects randomly assigned to this arm of the study will begin on active drug (100 mg BID bupropion) at week 1. At week 2, active drug is increased to 150mg BID unless subject reports one or more symptoms that are classified as moderate-severe. At week 4, subjects cross over to placebo for remainder of study. Subjects continue on placebo until end of study at week 8.
- Placebo-Bupropion: Subjects randomly assigned to this arm are given placebo at week 1. They will continue on placebo until week 4, at which time they will cross-over to bupropion 100 mg BID. At week 5, active drug is increased to 150mg BID unless subject reports one or more symptoms that are classified as moderate-severe. Subjects continue on active drug until end of study at week 8.
Arm/Group | Bupropion-Placebo | Placebo-Bupropion
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No